CLINICAL TRIAL: NCT02117778
Title: A Comparative Pulmonary Function Study of Continuous Supraclavicular, Suprascapular, and Interscalene Nerve Catheters After Total Shoulder Arthroplasty
Brief Title: Comparison of Pulmonary Function and Efficacy of Different Nerve Block Catheters for Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRI IRB13086
Record Dates: First submitted 2014-01-24; First posted 2014-04-21 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interscalene (Active Comparator): Continuous Interscalene Nerve Block
  Interventions: Procedure: Continuous Nerve Block
- Supraclavicular (Active Comparator): Continuous Supraclavicular Nerve Block
  Interventions: Procedure: Continuous Nerve Block
- Suprascapular (Active Comparator): Continuous Suprascapular Nerve Block
  Interventions: Procedure: Continuous Nerve Block

INTERVENTIONS:
Procedure: Continuous Nerve Block

SUMMARY:
This study is designed to evaluate lung function and pain control of continuous supraclavicular versus suprascapular versus interscalene nerve catheters in subjects undergoing total shoulder replacement. The investigators hypothesize that all three groups would have similar pain control; the supraclavicular and suprascapular groups may have better lung function.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral total shoulder arthroplasty
* ASA physical status I-III
* >18 years old
* Non-pregnant (or lactating)
* Consent to participate in the study

Exclusion Criteria:

* Refusal to participate
* < 18 years old
* Chronic opioid use
* Localized infection
* Pregnancy or lactating
* Pre-existing coagulopathy
* Allergy to ultrasound gel or local anesthetics
* Diaphragmatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Lung function | Post-Operative Day 1
  Vital Capacity, Spirometry

SECONDARY OUTCOMES:
Pain | Post Operative Day 1
  NRS Pain Scale
Opioid Consumption | Post Operative Day 1
  Total opioid consumption x 24 hours
Sensory and Motor Function | Post Operative Day 1
  Sensory Dermatome assessment C4 - C8 to touch; Motor assessment of grip and biceps with dynometer

CONTACTS AND LOCATIONS:
Overall Officials: David Auyong, MD, Principal Investigator — Physician
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States